CLINICAL TRIAL: NCT06617650
Title: GenerationGemelli: Longitudinal Study for the Evaluation of the Maternal Exposome on the Health of the Newborn and Child
Acronym: GenGem
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Boccia Stefania, Prof, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 4975
Record Dates: First submitted 2024-04-08; First posted 2024-09-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-04

CONDITIONS: Maternal Exposure; Maternal Exposure During Pregnancy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biological samples will be collected from both mothers and newborns (including vaginal swab, placenta sample, blood, saliva, meconium, and bronchoalveolar lavage fluid) at birth and within the early hours of the newborn's life.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The study involves the establishment of a case-control study within a birth cohort. With approximately 4,000 annual deliveries, the aim is to enroll 140 cases (newborns with intrauterine growth restriction [IUGR] and premature birth) and 280 controls each year, starting from September 2022. A comprehensive questionnaire will be utilized to gather information about various types of maternal environmental exposures before and during pregnancy. Biological samples will be collected from both mothers and newborns (including vaginal swab, placenta sample, blood, saliva, meconium, and bronchoalveolar lavage fluid) at birth and within the early hours of the newborn's life. Laboratory examinations will include the measurement of heavy metals and essential elements, investigation of placental distress and fetal brain damage biomarkers, analysis of microbiota, and assessment of DNA methylation profiles. Clinical follow-up assessments will be conducted in both cases and controls at 12 and 24 months, during which anthropometric data, types of feeding with particular reference to breastfeeding and its duration, pediatric emergency room visits, hospitalizations, medication usage, known allergies, and neuropsychological development will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Being resident for at least two years in the city of Rome, Italy.
* Being assisted and giving birth at FPG (presumably referring to a specific hospital).
* Meeting the definition of case or control.

Definitions:

- Cases:

Women with single pregnancies diagnosed with late intrauterine growth restriction (≥32 weeks of gestational age), according to the definition of Gordjin et al., in the absence of structural and/or evident organ malformations.

Women with spontaneous preterm birth at less than 32+0 weeks of gestational age.

- Controls:

Full-term pregnant women (gestational age between 37+0 and 41+6 weeks) without intrauterine growth restriction or other structural and/or genetic disorders.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants in the study will include all mother-child dyads classified as cases or controls who deliver at Fondazione Policlinico Gemelli (FPG). Out of 4,000 annual deliveries, an estimated 200 are classifiable as cases. Assuming a 70% response rate, it is anticipated that 140 cases and 280 controls will be enrolled per year, maintaining a 1:2 ratio. Enrollment will last for 24 months, with an expected total of 840 dyads. A missing rate of 20% is anticipated in the collection of biological samples due to lack of specific consent or logistical difficulties in obtaining samples at the time of enrollment.
Sampling Method: Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2022-09-15 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
To assess the association of individual exposures (and their interaction) with the incidence of high-risk pregnancy. | 2022-2024
  To assess the association of individual exposures (and their interaction) with the incidence of high-risk pregnancy.

CONTACTS AND LOCATIONS:
Locations (1):
- Dipartimento Universitario di Scienze della Vita e Sanità Pubblica, Roma, Italia, Italy